CLINICAL TRIAL: NCT02568696
Title: Activation of Coagulation Pathways in Clinical Renal Allotransplantation and Delayed Graft Function and Acute Rejection of the Graft
Brief Title: Intra-graft Coagulation Events in Clinical Renal Transplantation and Delayed Graft Function
Acronym: KTX
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: University of Helsinki (Other)
Responsible Party: Principal Investigator, Arie Passov, MD, Resident in Anaesthesiology and Intensive Care Medicine, Helsinki University Central Hospital
Other Study IDs: Dnro/64/13/03/02/2015; Dnro/64/13/03/02/2015 (Other: Ethics Committee, Department of Surgery, Hospital District of Helsinki and Uusimaa)
Record Dates: First submitted 2015-09-08; First posted 2015-10-06 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: End Stage Renal Disease; Reperfusion Injury; Delayed Graft Function; Kidney Transplantation
Keywords: kidney transplantation; renal transplantation; fibrinolysis; cell mediated rejection; coagulation; delayed graft function; Halloran criteria; graft rejection; thrombin generation; fibrin generation
MeSH Terms: conditions — Kidney Failure, Chronic; Reperfusion Injury; Delayed Graft Function; Thrombosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Three 4.5 ml citrated blood samples are taken during kidney transplantation surgery.
  Sample 1: taken after induction of anesthesia but before beginning of surgery from central venous catheter or by peripheral venous puncture.
  Sample 2 and 3: taken at 2 minutes after start of the reperfusion from the blood going into the transplant and the blood coming out of the transplant (iliac artery and renal vein respectively) by vessel puncture with a 24G needle. These samples are drawn into 5-ml syringes and transferred immediately into pyrogen free citrated vacuum tubes.
  Samples are centrifuged, plasma separated and divided into aliquots and stored at -80C.
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to investigate local activation of the coagulation system in the kidney graft during organ preservation and during early reperfusion in adult kidney transplantation. Generation of thrombin and fibrin as well as activation and inhibition of fibrinolysis will be investigated. Influence of these events on delayed graft function (DGF) and acute cell-mediated rejection will be evaluated.

DETAILED DESCRIPTION:
Background

In clinical kidney transplantation organ retrieval, cold-preservation of the graft as well as restoration of the blood flow to the transplant cause tissue damage (ischemia/reperfusion injury). Clinically these events can manifest themselves as delayed graft function (DGF), which is usually defined as the need for dialysis during first week after transplantation. DGF increases the risk of developing chronic rejection and subsequently loss of the transplant.

Ischaemia/reperfusion injury is biologically characterized by local profound inflammatory response, activation of the coagulation system and endothelial dysfunction in the transplanted organ. After reperfusion activated neutrophils cause tissue damage in the graft by production of reactive oxygen species (ROS) and release of proteolytic enzymes, which lead to plugging of the capillaries by accumulation of thrombocytes and fibrin. Blood flow is further diminished by increased blood viscosity and local vasoconstriction and swelling of the endothelial cells. Disorders of the microcirculation lead to "no-reflow" phenomenon whereby locally tissues remain ischemic, despite of good blood flow in the organ artery and vein.

Coagulation is activated in the renal transplant during reperfusion, when circulating factor VIIa (FVIIa) comes into contact with the tissue factor (TF), which is expressed on the endothelium due to ischaemia. FVII-TF complex activates factor X (FX) and activated FX (FXa) cleaves thrombin (FII) from prothrombin. Thrombin activates thrombocytes, cleaves fibrin from fibrinogen and activates factor XIII( FXIII), which stabilizes fibrin clot. Fibrin has been demonstrated to accumulate in the kidney graft during reperfusion. Fibrin accumulation is aggravated by inhibition of fibrinolysis due to reperfusion.

Furthermore, the investigators conducting this current research project, have previously gained indirect evidence in a small cohort study, that accumulation of fibrin occurs even before reperfusion, during donor care and organ retrieval. Most importantly, specifically this pre-reperfusion fibrin deposition was related to DGF.

Patients and sample size

There were several limitations in investigators previous study concerning intra-graft coagulation events in DGF. It was conducted as a part of a larger trial in renal transplantation and included only 30 patients in two study arms with different immunosuppressant regimens (peri-operative basiliximab and conventional triple therapy). Therefore, a new study, with larger sample size and standardized immunosuppression is warranted.

Therefore, in this current prospective observational study surgical technique, anaesthesia and hemodynamic management, immunosuppressive medications are strictly standardized. Sample size is increased to 100. The investigators prospectively screen all adult patients receiving their first kidney transplant from cadaveric donor. Only patients scheduled to receive local standard triple immunosuppressant therapy with cyclosporine A, mycophenolate mofetil and methylprednisolone are included.

Blood samples and prospective data collection

Blood samples for assessment of intra-graft coagulation events (generation of thrombin and fibrin, activation and inhibition of fibrinolysis) are drawn peri-operatively. Predefined clinical and demographical data are collected preoperatively and prospectively during 3 months after kidney transplantation to assess the influence of these coagulation events on delayed graft function according to Halloran criteria (8) (primary outcome) and acute cell mediated graft rejection (primary outcome).

ELIGIBILITY:
Inclusion Criteria:

* adult person (over 18 years old)
* cadaveric transplantation
* conventional standard immunosuppression plan (methylprednisolone, cyclosporin A, mycophenolate mofetil)

Exclusion Criteria:

* previous kidney transplant
* other than local standard immunosuppression
* panel reactive antibodies (PRA) >30%
* warfarin therapy
* dual anti-platelet therapy
* use of low molecular weight heparins (LMWH) or fondaparinux during last two weeks before surgery for other indication than hemodialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In Finland all adult kidney transplantation surgeries are performed at investigators institution. Study population consists of all adult patients fulfilling inclusion criteria admitted to the hospital for cadaveric renal transplantation.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-06; Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Trans-renal difference/ratio of plasma concentrations of coagulation measurements | Two minutes after reperfusion of the kidney transplant
  Trans-transplant difference/ratio is determined in order to correlate intra-graft coagulation events to the incidences of other primary outcomes.
Delayed Graft Function | During 1 week after kidney transplantation
  Delayed graft function is assessed by Halloran criteria: oliguria < 1000ml/24h for more than 2 days after transplantation or plasma creatinine >500 micromol/l during the first week after transplantation or more than one dialysis during the first week after transplantation (Halloran et al, Transplantation 1988;46:223-8.)
Acute cell mediated graft rejection | During 3 months after kidney transplantation

SECONDARY OUTCOMES:
Plasma creatinine value (micromol/L) | At admission to the hospital, during the first week after transplantation and at 1 and 3 months after renal transplantation
Plasma urea value (mmol/L) | At admission to the hospital, during the first week after transplantation and at 1 and 3 months after renal transplantation
Estimated glomerular filtration rate (ml/min/1.73 m2) | At admission to the hospital, during the first week after transplantation and at 1 and 3 months after renal transplantation
  Estimated glomerular filtration rate is calculated according to the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula
Urine output (ml/24h) | Pre-operative urine output (ml/24h) and daily urine output (ml/24h) during the first week after transplantation
  Urine output (ml/24h) before the surgery and during the first week after transplantation will be recorded
Renal artery and renal vein blood flow (ml/min) | Immediately after blood sample retrieval during reperfusion
  Renal artery and renal vein blood flow (ml/min) are measured intra-operatively immediately after blood sample retrieval using a specific probe
Fluid balance during surgery and post-anesthesia care unit stay (ml) | From the start of the kidney transplantation surgery until the discharge from post-anesthesia care unit (up to 24 hours from the start of the surgery)
  All fluids infused from the start of the kidney transplantation surgery until discharge from the post-anaesthesia care unit (until discharge to the ward) are recorded. All fluids losses (blood loss, urine output) during this period are recorded.
Transfusion | From the start of the kidney transplantation surgery until the discharge from post-anesthesia care unit (up to 24 hours from the start of the surgery)
  All blood products used during this time frame are recorded and reported
Prothrombin fragment 1+2 (F1+2) | Blood samples are taken at two timepoints: 1) immediately before the start of the surgery; 2) 2 minutes after reperfusion of the kidney transplant
  Preoperative value and the trans-transplant difference and/or ratio is determined in order to assess thrombin generation.
Fibrinopeptide A | Blood samples are taken at two timepoints: 1) immediately before the start of the surgery; 2) 2 minutes after reperfusion of the kidney transplant
  Preoperative value and the trans-transplant difference and/or ratio is determined in order to assess fibrin generation.
D-dimers | Blood samples are taken at two timepoints: 1) immediately before the start of the surgery; 2) 2 minutes after reperfusion of the kidney transplant
  Preoperative value and the trans-transplant difference and/or ratio is determined in order to assess fibrin degradation
Tissue type plasminogen activator | Blood samples are taken at two timepoints: 1) immediately before the start of the surgery; 2) 2 minutes after reperfusion of the kidney transplant
  Preoperative value and the trans-transplant difference and/or ratio is determined in order to assess activation of fibrinolysis.
Plasminogen activator inhibitor | Blood samples are taken at two timepoints: 1) immediately before the start of the surgery; 2) 2 minutes after reperfusion of the kidney transplant
  Preoperative value and the trans-transplant difference and/or ratio is determined in order to assess inhibition of fibrinolysis.
Syndecan-1 | Blood samples are taken at two timepoints: 1) immediately before the start of the surgery; 2) 2 minutes after reperfusion of the kidney transplant
  Preoperative value and the trans-transplant difference and/or ratio is determined in order to assess degradation of endothelial glycocalyx
Myeloperoxidase and/or lactoferrin | Blood samples are taken at two timepoints: 1) immediately before the start of the surgery; 2) 2 minutes after reperfusion of the kidney transplant
  Preoperative value and the trans-transplant difference and/or ratio is determined in order to assess activation of neutrophiles
Interleukin 6, interleukin 8, interleukin 10 | Blood samples are taken at two timepoints: 1) immediately before the start of the surgery; 2) 2 minutes after reperfusion of the kidney transplant
  Preoperative value and the trans-transplant difference and/or ratio is determined in order to assess activation/inhibition of inflammation
Number of hemodialyses and their indication after surgery | From the start of the surgery until 3 months after surgery
  All dialysis sessions will be recorded during first post-operative week. Indication for dialysis (oliguria, hyperkalemia, hypervolemia, acidosis) will be recorded during first post-operative week. At 1 and 3 months after surgery only number of dialyses/week will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Eero Pesonen, PhD, Study Chair — Helsinki University Central Hospital
Locations (1):
- Helsinki University and Helsinki University Hospital, Helsinki, Finland

REFERENCES:
- [Background] Eltzschig HK, Eckle T. Ischemia and reperfusion--from mechanism to translation. Nat Med. 2011 Nov 7;17(11):1391-401. doi: 10.1038/nm.2507. PMID 22064429
- [Background] Nemeth N, Furka I, Miko I. Hemorheological changes in ischemia-reperfusion: an overview on our experimental surgical data. Clin Hemorheol Microcirc. 2014;57(3):215-25. doi: 10.3233/CH-131648. PMID 23340000
- [Background] Sevastos J, Kennedy SE, Davis DR, Sam M, Peake PW, Charlesworth JA, Mackman N, Erlich JH. Tissue factor deficiency and PAR-1 deficiency are protective against renal ischemia reperfusion injury. Blood. 2007 Jan 15;109(2):577-83. doi: 10.1182/blood-2006-03-008870. Epub 2006 Sep 21. PMID 16990608
- [Background] Esmon CT. Targeting factor Xa and thrombin: impact on coagulation and beyond. Thromb Haemost. 2014 Apr 1;111(4):625-33. doi: 10.1160/TH13-09-0730. Epub 2013 Dec 12. PMID 24336942
- [Background] Sorensen-Zender I, Rong S, Susnik N, Lange J, Gueler F, Degen JL, Melk A, Haller H, Schmitt R. Role of fibrinogen in acute ischemic kidney injury. Am J Physiol Renal Physiol. 2013 Sep 1;305(5):F777-85. doi: 10.1152/ajprenal.00418.2012. Epub 2013 Jun 26. PMID 23804451
- [Background] Favreau F, Thuillier R, Cau J, Milin S, Manguy E, Mauco G, Zhu X, Lerman LO, Hauet T. Anti-thrombin therapy during warm ischemia and cold preservation prevents chronic kidney graft fibrosis in a DCD model. Am J Transplant. 2010 Jan;10(1):30-9. doi: 10.1111/j.1600-6143.2009.02924.x. Epub 2009 Dec 2. PMID 19958330
- [Background] Turunen AJ, Lindgren L, Salmela KT, Kyllonen LE, Petaja J, Pesonen EJ. Intragraft coagulation events and delayed graft function in clinical renal transplantation. Transplantation. 2008 Mar 15;85(5):693-9. doi: 10.1097/TP.0b013e31816615d8. PMID 18337662
- [Background] Halloran PF, Aprile MA, Farewell V, Ludwin D, Smith EK, Tsai SY, Bear RA, Cole EH, Fenton SS, Cattran DC. Early function as the principal correlate of graft survival. A multivariate analysis of 200 cadaveric renal transplants treated with a protocol incorporating antilymphocyte globulin and cyclosporine. Transplantation. 1988 Aug;46(2):223-8. PMID 3043779